CLINICAL TRIAL: NCT01411683
Title: Mandibular Overdentures Retained by Conventional or Mini Implants: a Randomized Clinical Trial
Brief Title: Mandibular Overdentures Retained by Conventional or Mini Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Raphael Freitas de Souza, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FORP-PT-004; 2011.1.197.58.3 (Other: Institutional Review Board (FORP-USP)); 2011/00688-7 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Edentulous Mouth; Edentulous Jaw
Keywords: Cost estimates; Complete Denture; Dental Economics; Dental Implants; Dental Prosthesis, Implant-Supported; Denture Retention; Edentulous; Edentulism; Mini dental implant; Oral Health-Related Quality of Life; Overdenture; Patient Acceptance of Health Care; Quality of Health Care; Quality of Life; Patient Satisfaction
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous; Patient Acceptance of Health Care; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 mini dental implants (Experimental): Retention of an overdenture by means of 4 mini implants.
  Interventions: Device: Implant-retained mandibular overdenture
- 2 mini dental implants (Experimental): Retention of an overdenture by means of 2 mini implants.
  Interventions: Device: Implant-retained mandibular overdenture
- 2 conventional dental implants (Active Comparator): Retention of an overdenture by means of 2 conventional implants associated to ball attachments.
  Interventions: Device: Implant-retained mandibular overdenture

INTERVENTIONS:
Device: Implant-retained mandibular overdenture — Insertion of implants in the lower arch in order to retain existing complete dentures. Tested implants are approved by the Brazilian National Health Surveillance Agency for clinical use.
  Other Names: - Mini-implant overdenture.

SUMMARY:
This study aims to compare mandibular overdentures retained either by mini or standard size implants as a treatment for edentulous adults, in terms of patient-reported satisfaction and oral health-related quality of life. We will also evaluate post surgical discomfort, the success rate of prostheses and implants in the long term, denture quality and costs.

ELIGIBILITY:
Inclusion Criteria:

* Complete edentulism;
* Request of implant stabilization of the existing lower conventional denture;
* Clinically acceptable maxillary and mandibular complete dentures;
* Adequate space in the anterior mandible for the placement of four mini implants and two conventional implants (regular diameter);
* Ability to maintain adequate oral hygiene and clean dentures;
* Systemic health status that permits minor surgical procedures;
* Adequate understanding of written and spoken Portuguese;
* Capacity of giving written informed consent.

Exclusion Criteria:

* Lack of minimum vertical mandibular bone height of 11mm in the interforaminal region;
* Acute or chronic symptoms of parafunctional disorders;
* History of radiation therapy to the orofacial region;
* Specific conditions that may jeopardize the treatment, i.e. alcoholism and smoking;
* Severe/serious illness that requires frequent hospitalization;
* Impaired cognitive function;
* Impossibility to return for evaluations/study recalls.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Denture satisfaction | 2 years
  To be assessed by specific questionnaires
Oral health-related quality of life | 2 years
  To be assessed by means of the Brazilian version of the OHIP-EDENT.

SECONDARY OUTCOMES:
Post-surgical discomfort | 7 days
  Pain and discomfort following the insertion of dental implants, as assessed by a specific questionnaire.
Success rate of implant-retained mandibular overdentures | 2 years
  Survival of implant-retained overdentures.
Denture quality | 2 years
  Functional aspects of mandibular overdentures, as assessed by a dentist.
Treatment costs | 2 years
  This outcome will be measured by means of specific forms, according to 2 components:
  * Direct costs: cost of labor, materials, radiographs and medications;
  * Indirect costs: patient's time and transportation expenses.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael F de Souza, DDS, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Ribeirão Preto Dental School, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chaves CA, Souza RF, Cunha TR, Vecchia MP, Ribeiro AB, Bruniera JF, Silva-Sousa YT. Preliminary In Vitro Study on O-Ring Wear in Mini-Implant-Retained Overdentures. Int J Prosthodont. 2016 Jul-Aug;29(4):357-9. doi: 10.11607/ijp.4677. PMID 27479342
- [Result] Ribeiro AB, Della Vecchia MP, Cunha TR, Sorgini DB, Dos Reis AC, Muglia VA, de Albuquerque RF Jr, de Souza RF. Short-term post-operative pain and discomfort following insertion of mini-implants for retaining mandibular overdentures: a randomized controlled trial. J Oral Rehabil. 2015 Aug;42(8):605-14. doi: 10.1111/joor.12287. Epub 2015 Mar 13. PMID 25765784
- [Result] de Souza RF, Ribeiro AB, Della Vecchia MP, Costa L, Cunha TR, Reis AC, Albuquerque RF Jr. Mini vs. Standard Implants for Mandibular Overdentures: A Randomized Trial. J Dent Res. 2015 Oct;94(10):1376-84. doi: 10.1177/0022034515601959. Epub 2015 Aug 20. PMID 26294416
- [Result] dos Reis AC, Leon JE, Ribeiro AB, Della Vecchia MP, Cunha TR, de Souza RF. Traumatic ulcerative granuloma with stromal eosinophilia around mini dental implants without the protection of a denture base. J Prosthodont. 2015 Jan;24(1):83-6. doi: 10.1111/jopr.12184. Epub 2014 Jun 27. PMID 24975725
- [Derived] Della Vecchia MP, Leles CR, Cunha TR, Ribeiro AB, Sorgini DB, Muglia VA, Reis AC, Albuquerque RF Jr, de Souza RF. Mini-Implants for Mandibular Overdentures: Cost-Effectiveness Analysis alongside a Randomized Trial. JDR Clin Trans Res. 2018 Jan;3(1):47-56. doi: 10.1177/2380084417741446. Epub 2017 Nov 20. PMID 30938654
- See also: Institutional page of the Ribeirão Preto Dental School (research site) — http://www.forp.usp.br
- See also: Principal Investigator´s CV (RF de Souza) — http://lattes.cnpq.br/7092555880664311
- See also: Principal Investigator´s CV (RF Albuquerque Jr) — http://lattes.cnpq.br/5953029548378417